CLINICAL TRIAL: NCT06818682
Title: Reduced Length of ADT and ARTA With XRT in High-Risk Prostate Cancer (RELAX): A Randomised Trial
Acronym: RELAX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Vedang Murthy, Professor, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 901060
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Prostate Carcinoma
Keywords: Prostate Cancer; Prostate Radiotherapy; Hormone therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Arm (Experimental): Radiotherapy to prostate and pelvic nodes (66-68Gy and 50Gy in 25 fractions OR 60-62Gy and 44Gy in 20 fractions OR 36.25-40Gy and 25Gy in 5 fractions) with ADT for 9 months and ARTA for 6 months
  Interventions: Drug: ADT for 9 months and ARTA for 6 months
- Standard Arm (Active Comparator): Radiotherapy to prostate and pelvic nodes (66-68Gy and 50Gy in 25 fractions OR 60-62Gy and 44Gy in 20 fractions OR 36.25-40Gy and 25Gy in 5 fractions) with ADT for 2 years
  Interventions: Drug: ADT for 2 years

INTERVENTIONS:
Drug: ADT for 9 months and ARTA for 6 months — Radiotherapy to prostate and pelvic nodes (66-68Gy and 50Gy in 25 fractions OR 60-62Gy and 44Gy in 20 fractions OR 36.25-40Gy and 25Gy in 5 fractions) with ADT for 9 months and ARTA for 6 months
  Arms: Test Arm
Drug: ADT for 2 years — Radiotherapy to prostate and pelvic nodes (66-68Gy and 50Gy in 25 fractions OR 60-62Gy and 44Gy in 20 fractions OR 36.25-40Gy and 25Gy in 5 fractions) with ADT for 2 years
  Arms: Standard Arm

SUMMARY:
Aim of the study to improve the treatment of high-risk non-metastatic prostate cancer by comparing reduced duration of hormone therapy to the standard duration of two years, when combined with curative intent standard of care radiotherapy to prostate and pelvic nodes. The reduced duration will be intensified with addition of newer hormonal agents such as abiraterone or enzalutamide tablets, which have been shown to improve disease control in locally advanced prostate cancer. This is hoped to reduce the side effects of prolonged hormone therapy, while maintaining similar rates of disease control and survival.

The effectiveness of both treatment approaches will be assessed in terms of cancer control, survival, and overall quality of life of patients. Additionally, the study will examine the side effects associated with each treatment regimen, which could provide valuable insights into impact of treatment duration on patients. If a person decides not to participate, they will still receive the standard two years of hormonal therapy and radiation therapy outside the study. This ensures that all patients receive appropriate care regardless of their involvement in the research. Participation is voluntary, and will not affect patient care.

ELIGIBILITY:
Inclusion Criteria:-

* Patients with biopsy proven prostate adenocarcinoma, deemed suitable for curative- intent radiotherapy
* Clinicoradiological stage T1-T4N0M0 using PSMA-PETCT and MRI
* High risk or very high risk (as per NCCN 2023): stage T3a + OR Gleason Score 4+4 or 4+5 OR PSA 20 +
* Patient fit and able to receive ADT for 2 years
* Patient fit and able to receive ARTA for 6 months
* ECOG performance status 0-2
* Patient able and willing for informed consent and reliable for follow-up

Exclusion Criteria:-

* Primary Gleason pattern 5 (Gleason score 5+4 or 5+5)
* Life expectancy deemed to be less than 2 years
* Uncontrolled comorbidities such as diabetes or hypertension causing ineligibility to receive ARTA
* Bulky primary disease with extensive infiltration into bladder/rectum/pelvic muscle
* Prior ADT more than 3 months before screening or prior orchiectomy
* Prior prostatectomy
* Unsuitable for curative dose of radiotherapy (severe urinary obstructive symptoms, inflammatory bowel disease, prior pelvic radiotherapy etc.)
* Presence of adverse pathological variants (such as small cell histology)
* Unable or unwilling to consent and follow up

Ages: 19 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS), defined as the time to first clinicoradiological recurrence or death due to any cause, from the date of randomisation. | 5 years

SECONDARY OUTCOMES:
Biochemical failure free survival (BFFS) | 5-year
  Time to biochemical failure (nadir PSA + 2ng/mL) or death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
May be shared request of PI